CLINICAL TRIAL: NCT00079235
Title: A Phase II Study of the mTOR Inhibitor, CCI-779 in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: CCI-779 in Treating Patients With Stage IIIB (With Pleural Effusion) or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01810; N0323; CDR0000355117; NCCTG-N0323; U10CA025224 (NIH)
Record Dates: First submitted 2004-03-08; First posted 2004-03-10 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-06

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — temsirolimus; Sirolimus

ARMS (1):
- Arm I (Experimental): Patients receive CCI-779 IV over 30 minutes on days 1, 8, 15, and 22.
  Interventions: Drug: temsirolimus; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: temsirolimus — Given IV
  Other Names: CCI-779; cell cycle inhibitor 779; Torisel
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well CCI-779 works in treating patients with stage IIIB non small cell lung cancer (with pleural effusion) or stage IV non-small cell lung cancer. Drugs used in chemotherapy, such as CCI-779, work in different ways to stop tumor cells from dividing so they stop growing or die. CCI-779 may also stop the growth of tumor cells by blocking the enzymes necessary for their growth.

DETAILED DESCRIPTION:
OBJECTIVES: Primary I. Determine the response rate in patients with stage IIIB (with pleural effusion) or IV non-small cell lung cancer treated with CCI-779.

II. Determine the clinical toxic effects of this drug in these patients.

Secondary I. Determine the 24-week progression-free survival rate in patients treated with this drug.

II. Determine the time to progression and overall survival of patients treated with this drug.

III. Evaluate predictive markers of activity (e.g., PTEN mutations and phosphoAkt expression) of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive CCI-779 IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 6 months for up to 5 years.

PROJECTED ACCRUAL: A total of 25-55 patients will be accrued for this study within 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)

  * Stage IIIB (with pleural effusion) or IV disease
* Measurable disease

  * At least 1 lesion ≥ 2.0 cm by conventional techniques OR ≥ 1.0 cm by spiral CT scan
  * The following are not considered measurable disease:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Inflammatory breast disease
    * Lymphangitis cutis/pulmonis
    * Cystic lesions
    * Abdominal masses that are not confirmed and followed by imaging techniques
* Blood and tissue blocks available
* Must have accessible tumor (i.e., superficial lesions such as lymph node, subcutaneous nodules) to provide core needle biopsy tissue before and during study treatment
* No known brain metastases
* Performance status - ECOG 0-2
* At least 12 weeks
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL
* Bilirubin ≤ 2 times upper limit of normal (ULN)
* AST ≤ 3 times ULN (5 times ULN if hepatic metastases are present)
* Creatinine ≤ 1.5 times ULN
* Serum fasting cholesterol ≤ 350 mg/dL
* Serum fasting triglycerides ≤ 400 mg/dL
* HIV negative
* No uncontrolled infection
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or non-invasive carcinomas
* No concurrent severe underlying disease that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study treatment
* No prior biologic therapy
* No prior gene therapy
* No prior immunotherapy
* No concurrent immunotherapy
* No concurrent prophylactic growth factors to support neutrophil count
* No prior chemotherapy for NSCLC except low-dose cisplatin as a radiosensitizer
* No other concurrent chemotherapy
* No concurrent dexamethasone (10 mg IV)
* No prior radiotherapy to 30% or more of bone marrow
* Concurrent radiotherapy for underlying malignancy and non-target sites (e.g., painful pre-existing bony metastasis) allowed
* No other concurrent investigational therapy
* No concurrent immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-02; Primary Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Confirmed tumor response according to the Response Evaluation Criteria in Solid Tumors (RECIST) | Up to 5 years
  Confidence intervals for the true success proportion will be calculated using the Duffy-Santner approach.

SECONDARY OUTCOMES:
Progression-free survival | 24 weeks
  Computed and binomial confidence intervals for the true success proportion will be calculated.
Survival time | Time from registration to death due to any cause, assessed up to 5 years
  Estimated using the method of Kaplan-Meier.
Time to disease progression | Time from registration to documentation of disease progression, assessed up to 5 years
  Estimated using the method of Kaplan-Meier.
Effects of CCI-779 on mTOR as assessed by expression of 4EBP, phosphoAkt, p70S6kinase, eIF4E, cyclinD1, Her2, and EGFR | Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Alex Adjei, Principal Investigator — North Central Cancer Treatment Group
Locations (1):
- North Central Cancer Treatment Group, Rochester, Minnesota, United States